CLINICAL TRIAL: NCT01306526
Title: Intravascular Ultrasound Diagnostic Evaluation of Atherosclerosis in Singapore- Obstructive Sleep Apnea (IDEAS-OSA) Study
Brief Title: Relationship Between Obstructive Sleep Apnea and Coronary Atherosclerosis
Acronym: IDEAS-OSA
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Chi-Hang Lee, Associate Professor, National University of Singapore
Other Study IDs: DSRB: C/10/341
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease; Obstructive Sleep Apnea
Keywords: Thin-cap fibroatheroma; Vulnerable plaque; Coronary artery disease; Obstructive sleep apnea; Intravascular Ultrasound
MeSH Terms: conditions — Coronary Artery Disease; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate to Severe OSA

SUMMARY:
Obstructive sleep apnea (OSA) is a respiratory disorder of sleep characterized by recurrent episodes of complete or partial upper airway obstruction, leading to intermittent oxygen deprivation. This results in sympathetic activation and surges in blood pressure, production of vasoactive substances, as well as activation of the inflammatory and procoagulant pathways. Epidemiological evidence indicates the prevalence of OSA is higher in patients with coronary artery disease than in the general population. The investigators recently showed that 65.7% and 41.9% of the Singapore patients admitted with myocardial infarction were found to have previously undiagnosed OSA and severe OSA, respectively. In a 10-year follow-up epidemiological study, OSA was independently associated with a higher prevalence of fatal and non-fatal cardiovascular events among the otherwise healthy general population. The investigators further showed that in patients who have undergone primary percutaneous coronary intervention for acute myocardial infarction, OSA was an independent predictor of future adverse event rates. Despite the observed association between OSA and adverse cardiovascular outcomes, the underlying pathophysiological mechanisms remain unclear. In this proposal, the investigators aim to elucidate the relationship between OSA and composition of coronary atherosclerotic plaques.

ELIGIBILITY:
Inclusion Criteria:

* Angiogrqaphically documented coronary artery disease
* De novo lesion
* Native coronary artery

Exclusion Criteria:

* known OSA
* intubation and mechanical ventilation
* electrical instability with a high risk of malignant ventricular arrhythmia
* cardiogenic shock
* previous coronary artery bypass surgery
* chronic renal failure on dialysis
* inability to give informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 21 to 80 years who are scheduled to undergo either an elective, urgent or emergent diagnostic coronary angiography are eligible
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Total Atheroma Volume | Baseline
  Relationship between OSA and Total Atheroma Volume determined (IVUS) will be determined

SECONDARY OUTCOMES:
Thin-cap fibroatheroma | Baseline
  Relation between OSA and prevalence of thin-cap fibroatheroma (VH-IVUS) will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- National University Health System, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Lee CH, Sethi R, Li R, Ho HH, Hein T, Jim MH, Loo G, Koo CY, Gao XF, Chandra S, Yang XX, Furlan SF, Ge Z, Mundhekar A, Zhang WW, Uchoa CH, Kharwar RB, Chan PF, Chen SL, Chan MY, Richards AM, Tan HC, Ong TH, Roldan G, Tai BC, Drager LF, Zhang JJ. Obstructive Sleep Apnea and Cardiovascular Events After Percutaneous Coronary Intervention. Circulation. 2016 May 24;133(21):2008-17. doi: 10.1161/CIRCULATIONAHA.115.019392. Epub 2016 May 13. PMID 27178625
- [Derived] Tan A, Hau W, Ho HH, Ghaem Maralani H, Loo G, Khoo SM, Tai BC, Richards AM, Ong P, Lee CH. OSA and coronary plaque characteristics. Chest. 2014 Feb;145(2):322-330. doi: 10.1378/chest.13-1163. PMID 24178625